CLINICAL TRIAL: NCT03407872
Title: One-centre Safety and Pharmacokinetics Phase I Study of Inhaled Esketamine in Healthy Volunteers With Two Single Ascending Dose and One Double-blind Multiple Ascending Dose Parts
Brief Title: Safety and Pharmacokinetic Study of Inhaled Esketamine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 01KET2017
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Only PART C will be double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PART A (Experimental): 6 cohorts will receive single dose of Esketamine DPI administered with dose escalation between cohorts.
  Interventions: Drug: Esketamine DPI
- PART B (Experimental): 4 cohorts will receive single dose of Esketamine DPI administered with dose escalation between cohorts.
  Interventions: Drug: Esketamine DPI
- PART C (Experimental): 4 cohorts will receive multiple dose of Esketamine DPI in two weeks' time administered with dose escalation between cohorts.
  Interventions: Drug: Esketamine DPI
- PART C placebo (Placebo Comparator): 4 cohorts will receive multiple dose of matching placebo in two weeks' time.
  Interventions: Drug: Placebo DPI

INTERVENTIONS:
Drug: Esketamine DPI — Participants will receive different number of consecutive Esketamine DPI inhalations, consider as a single dose. There will be dose escalation between cohorts.
  Arms: PART A
Drug: Esketamine DPI — Participants will receive different dosing sequences of Esketamine DPI inhalations, consider as a single dose. There will be dose escalation between cohorts. Number of Esketamine DPI inhalations within a dosing sequence will be defined based on results from PART A of the study.
  Dose: very low, low, medium, high.
  Arms: PART B
Drug: Esketamine DPI — Participants will receive different cycle of treatment consisting of 4 dosing sequences administered within 2 weeks. There will be dose escalation between cohorts. Participants in this part will be randomized to receive Esketamine DPI or placebo in 3:1 ratio. Number of Esketamine DPI inhalations within a dosing sequence will be defined based on results from PART A and PART B of the study.
  Dose: very low, low, medium, high.
  Arms: PART C
Drug: Placebo DPI — Participants will receive different cycle of treatment consisting of 4 dosing sequences administered within 2 weeks. Participants in this part will be randomized to receive Esketamine DPI or placebo in 3:1 ratio.
  In each cohort, number of placebo inhalations within a dosing sequence will correspond to number of Esketamine DPI inhalations.
  Arms: PART C placebo

SUMMARY:
The planned study is to determine the pharmacokinetic properties of Esketamine and safety assessment with inhaled Esketamine after different number of inhalations and different dosing sequences within three parts of the study.

DETAILED DESCRIPTION:
This is to be one-centre, single ascending dose and double-blind placebo controlled multiple dose three part study of Esketamine DPI (dry powder inhaler) in healthy volunteers.

PART A is a single dose, open-label part with Esketamine DPI inhalations administered with dose escalation between cohorts.

PART B is a single dose, open-label part with Esketamine DPI inhalations administered in different dosing sequences with dose escalation between cohorts.

PART C is a multiple dose, double-blind, placebo-controlled part with Esketamine DPI inhalations administered in different cycles of treatment (with four dosing sequences within two weeks) with dose escalation between cohorts. Participants in this part will be randomized to receive Esketamine DPI or placebo in 3:1 ratio.

Pharmacokinetic properties and safety of Esketamine DPI will be determined following different number of inhalations in PART A, different dosing sequences in PART B and different cycles of treatment in PART C.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian female or male,
* Age: 18-55 years old, inclusive,
* Body-mass index (BMI): ≥18.5 kg/m^2 and <29.9 kg/m^2
* Non-smoker and nonuser of tobacco products for at least 1 year before screening,
* Physical examination without any clinically relevant abnormality,
* Laboratory values not clinically significant,
* Volunteer (or his/her partner) of childbearing potential willingness to use acceptable forms of contraception.

Exclusion Criteria:

* Known allergy or hypersensitivity to ketamine or its derivates and/or to any study product excipients,
* Any known significant current or past acute or chronic disease or condition,
* Participation in other clinical trial within 90 days preceding the screening,
* Blood drawn within 30 days prior to inclusion to the study (more or equal to 300mL),
* Positive results from pregnancy test for female participants,
* Lactation in women participants,
* Hypotension or hypertension in medical history,
* Narcotic, alcohol addiction or abuse,
* Participant who adhere to a special diet (e.g. low calories, vegetarian).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-12-09 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Cmax - maximum Esketamine plasma concentration | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The maximum concentration of the Esketamine in plasma after drug administration, obtained directly from the measured concentrations.
AUC (0-24) - area under the Esketamine plasma concentration-time curve from time 0 to 24 hours after study drug administration | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The AUC(0-24) is a measure of total plasma exposure to the drug from time point zero to 24 hours after study drug administration.
Number of inhalations needed to achieve the assumed Esketamine antidepressive plasma concentration. | up to 24 hours after study drug administration in PART A
Number of inhalations within dosing sequence needed to maintain the assumed Esketamine antidepressive plasma concentration. | up to 24 hours after study drug administration in PART B

SECONDARY OUTCOMES:
AUC (0-inf) - area under the Esketamine plasma concentration-time curve from time 0 to infinity time | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The AUC(0-inf) is a measure of total plasma exposure to the drug from time point zero extrapolated to infinity.
Tmax - time to reach maximum Esketamine plasma concentration | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The Tmax is time to reach the maximum plasma concentration (Cmax), obtained directly from the actual sampling times.
Kel -elimination rate constant | up to 24 hours after each study drug administration in PART A, B and C of the study.
  Kel will be estimated via linear regression of time versus log of concentration.
T1/2 - plasma elimination half-life for Esketamine | up to 24 hours after each study drug administration in PART A, B and C of the study.
  T1/2 will be calculated as 0.693/Kel.
Cmax - maximum Esnorketamine plasma concentration | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The maximum concentration of the Esnorketamine in plasma after drug administration, obtained directly from the measured concentrations. Esnorketamine is Esketamine's main metabolite.
AUC (0-24) - area under the Esnorketamine plasma concentration-time curve from time 0 to 24 hours after study drug administration. | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The AUC(0-24) is a measure of total Esnorketamine plasma exposure to the metabolite from time point zero to 24 hours after study drug administration. Esnorketamine is Esketamine's main metabolite.
Tmax - time to reach maximum Esnorketamine plasma concentration. | up to 24 hours after each study drug administration in PART A, B and C of the study.
  The Tmax is time to reach the maximum Esnorketamine plasma concentration (Cmax), obtained directly from the actual sampling times. Esnorketamine is Esketamine's main metabolite.
Number of participants with adverse events (AEs) and Serious Adverse Events (SAEs). | up to 7 days in PART A and PART B of the study and up to 25 days in PART C of the study.
  Participants during hospitalization will be closely observed to assure maximal safety and to collect occurrence of all adverse event. To follow-up on all study participants telephone calls with a request for information regarding their health condition will be made. All adverse events will be collected with special attention to occurrence of psychotomimetic and dissociative effects after study drug administration.

CONTACTS AND LOCATIONS:
Locations (1):
- BioResearch Group Sp. z o.o., Kajetany, Poland

IPD SHARING:
Plan to Share IPD: No